CLINICAL TRIAL: NCT05557110
Title: A Multicenter, Single-arm, Open-end Study of Reduced-dose Chemotherapy Followed by Blinatumomab in Induction Therapy of Newly Diagnosed Non-elderly Philadelphia Chromosome Negative Acute B Lymphoblastic Leukemia
Brief Title: Reduced-dose Chemotherapy Followed by Blinatumomab in Induction Therapy of Newly Diagnosed Non-elderly Ph-B-ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chen Suning (Other)
Responsible Party: Sponsor-Investigator, Chen Suning, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ALL02
Record Dates: First submitted 2022-09-16; First posted 2022-09-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: B Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; Ph-B-ALL; Induction therapy
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- reduced-intensity chemotherapy followed by berintuzumab (Experimental): Induction therapy was performed with reduced intensity chemotherapy (including 1 dose of Idarubicin 8 mg/m2, 1 dose of Vindesine 3 mg/m2, and 7 days of Dexamethasone 9 mg/m2/d) followed by 2 weeks of Blinatumomab (9 ug/d d8-14, 28 ug/d d15-21) immediately. Bone marrow evaluation was performed on day 22±2, and consolidation therapy was performed after achieving bone marrow remission (CR/CRh/CRi). If CR/CRh/CRi was not achieved in the first course of induction therapy, Blinatumomab (28ug/d×14d) should be continued and bone marrow evaluation should be evaluated again.
  The regimen of consolidation therapy is recommended as multidrug combination chemotherapy (including high-dose Methotrexate or Cytarabine combined with Asparaginase) or alternating with Blinatumomab (28 ug/d×28d). If Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT) is not performed, consolidation therapy needs at least 4 courses before 2 years maintenance therapy.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Reduced-intensity chemotherapy followed by Blinatumomab

SUMMARY:
Blinatumomab, a CD3/CD19 bisespecific T-cell conjugative antibody, has shown high efficacy in phase I/II studies of relapsed/refractory B-lymphoblastic leukemia (B-ALL), particularly in the context of low tumor burden.Meanwhile, Blinatumomab also plays an important role in rapid and efficient clearance of MRD in patients. Therefore, its use in combination with less intensive chemotherapy for initial induction therapy in newly diagnosed patients may result in favorable response rates, greater depth of remission, and lower treatment-related toxic effects.

In this study, newly diagnosed non-elderly patients with Philadelphia chromosomal negative (PH-) B-ALL were enrolled and treated with reduced-intensity chemotherapy followed by Blinatumomab as the basis of induction therapy. The clinical remission rate, MRD negative rate and treaty-related adverse reactions were evaluated in newly diagnosed non-elderly PH-B-ALL patients during induction therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-65
2. Ph-(BCR-ABL1 negative)B-ALL was diagnosed according to WHO diagnostic criteria
3. Newly diagnosed patients without prior induction therapy (except hydroxyurea and glucocorticoids ≦5 days)
4. ECOG score 0-3
5. Liver function: total bilirubin ≦ 3 times the upper limit of normal; Alanine aminotransferase ≦ 3 times upper limit of normal motion; Aspartate aminotransferase ≦ 3 times upper limit of normal motion; (except considering leukemia infiltration)
6. Renal function: endogenous creatinine clearance ≧30ml/min
7. Patients must be able to understand and willing to participate in the study and must sign the informed consent form.

Exclusion Criteria:

1. Ph+ (BCR-ABL1 positive) ALL and known ABL class Ph-Like ALL
2. T cells ALL
3. Mature B-cell leukemia/lymphoma, B-cell lymphoma, isolated extramedullary disease
4. Acute mixed-cell leukemia
5. Central nervous system leukemia
6. HIV infection
7. HBV-DNA or HCV-RNA positive
8. Patients with grade 2 or higher heart failure and other patients deemed inappropriate for inclusion by the investigator
9. Pregnant or breastfeeding patients
10. The study patient was refused enrollment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Induction therapy phase: The time of bone marrow evaluation is day 22 or 37±2.
  Overall response rate (ORR), including complete response (CR)/ complete response rate with partial hematologic recovery (CRh)/ complete response rate with incomplete hematologic recovery (CRi).

SECONDARY OUTCOMES:
The negative rate of minimal residual lesion (MRD) | Induction therapy phase: The time of bone marrow evaluation is day 22 or 37±2.
  The negative rate of minimal residual lesion (MRD) during induction therapy (The threshold is 1×10^-4)
Treatment-related SAE | From the beginning of induction therapy to the beginning of consolidation therapy.
  Incidence of treatment-related severe adverse events, including severe bleeding, infection, drug-related adverse events, and organ dysfunction.
Time of hematopoietic recovery | From the beginning of induction therapy to the beginning of consolidation therapy.
  The duration of the patient in the granulocytic deficiency and thrombocytopenia phases.
Event-free survival (EFS) | 1 year after study completion
  The time from enrollment to the occurrence of any event, including death, progression of disease, change in treatment regimen, and occurrence of fatal or intolerable side effects.
Overall survival (OS) | 1 year after study completion
  From the time of enrollment in the study to the time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, PHD, Principal Investigator — The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lu J, Qiu H, Wang Y, Zhou X, Dai H, Lu X, Yang X, Gu B, Hong M, Miao M, Lu R, Wang J, Wu Q, Xue M, Wang Y, Deng A, Shen Y, Liu Y, Dou X, Lei Y, Wu D, Zhu Y, Chen S. Reduced-dose chemotherapy and blinatumomab as induction treatment for newly diagnosed Ph-negative B-cell precursor acute lymphoblastic leukemia: a phase 2 trial. J Hematol Oncol. 2024 Sep 2;17(1):79. doi: 10.1186/s13045-024-01597-8. PMID 39218935
- [Derived] Lu J, Zhu Y, Qiu H, Wang Y, Zhou X, Dai H, Lu X, Gu B, Hong M, Miao M, Lu R, Wang J, Wu Q, Xue M, Wang Y, Deng A, Shen Y, Liu Y, Dou X, Lei Y, Yang X, Chen S. Reduced-dose chemotherapy followed by blinatumomab for newly diagnosed philadelphia chromosome-negative B-cell precursor acute lymphoblastic leukemia: a propensity-matched comparison with hyper-CVAD. Discov Oncol. 2025 Feb 21;16(1):223. doi: 10.1007/s12672-025-01968-8. PMID 39984805
- See also: 2024EHA; P409 — http://library.ehaweb.org/eha/2024/eha2024-congress/420473/jing.lu.blinatumomab.induction.therapy.following.reduced-dose.chemotherapy.in.html?f=listing%3D4%2Abrowseby%3D8%2Asortby%3D2%2Amedia%3D3%2Aspeaker%3D1000669